CLINICAL TRIAL: NCT07276243
Title: Comparação da eficácia clínica e estética Entre o Tratamento de Varizes Com Espuma de Polidocanol Associada ou não ao Laser transdérmico: Ensaio clínico Randomizado
Brief Title: Polidocanol Foam With or Without Transdermal Laser for Varicose Veins: Randomized Clinical Trial
Acronym: POLI-LASER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Pedro Ernesto (Other)
Responsible Party: Principal Investigator, Juliana de Miranda Vieira, Principal Investigator, Hospital Universitario Pedro Ernesto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUPE-Varizes-Laser-2026
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will be performed in a 1:1 ration using a concealed allocation sequence accessible only at the time of treatment by a staff member not involved in outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Foam only (Active Comparator): Polidocanol 0,5% foam prepared with 1 mL of sclerosant and 3 mL of room air, injected under visualization of reticular vein (5 - 8 mL total).
  Interventions: Drug: Polidocanol foam sclerotherapy
- Group B: Foam + Laser (Experimental): Polidocanol 0,25% foam (1 mL of sclerosant + 2 mL of room air) followed within 2 minutes by long-pulse Nd:YAG 1064 nm laser (spot 6 mm; pulse 20-30 ms; fluence 60-70 J/cm²), with skin cooling.
  Interventions: Drug: Polidocanol foam sclerotherapy; Device: Transdermal Nd:YAG 1064 nm laser

INTERVENTIONS:
Drug: Polidocanol foam sclerotherapy — Polidocanol foam prepared using the Tessari method. Concentration 0,5% (Foam Arm) or 0,25% (Foam + Laser Arm), injected under ultrasound guidance.
Device: Transdermal Nd:YAG 1064 nm laser — Long-pulse Nd:YAG 1064 nm transdermal laser applied along the treated vein path immediately after foam injection.
  Arms: Group B: Foam + Laser

SUMMARY:
This randomized, double-blind, parallel clinical trial will compare the clinical and aesthetic outcomes of polidocanol foam sclerotherapy alone versus polidocanol foam associated with long-pulse 1064 nm Nd:YAG transdermal laser in the treatment of lower limb tributary varicose veins. The primary endpoint is venous occlusion rate at 30 days assessed by Doppler ultrasound. Secondary outcomes include cutaneous hyperpigmentation, pain, patient satisfaction, and adverse events.

DETAILED DESCRIPTION:
The study aims to evaluate whether the association of transdermal Nd:YAG 1064 nm laser with polidocanol foam improves venous occlusion and aesthetic outcomes compared to foam alone. Participants will be adult patients with lower limb varicose veins CEAP 1-3 confirmed by Doppler ultrasound. After randomization (1:1), the control group will receive 0.5% polidocanol foam, while the intervention group will receive 0.25% polidocanol foam followed by transdermal laser application. A second session will be performed only if partial occlusion persists at the 30-day follow-up. Assessments will include venous occlusion at 30, 90 and 180 days after the procedure, pigmentation, pain intensity, number of sessions required, patient satisfaction, and adverse events. Standardized photographs will be taken at baseline, 30, 90 and 180 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 75 years
* CEAP clinical class 1-3
* Lower limb tributary varicose veins 2,5 to 4,0 mm in diameter on Doppler ultrasound.
* Vein depth up to 4 mm from the skin surface.
* Tributary vein may originate from the great or samll saphenous vein as long as the saphenous vein is competent on Doppler.
* Reflux limited to the target tributary.
* Body mass index (BMI) < 35 km/m²
* Able and willing to provide informed consent.

Exclusion Criteria:

* CEAP clinical class ≥ 4
* Axial reflux of the great or small saphenous vein requiring prior treatment
* Tributary vein diameter < 2.5 mm or > 4.0 mm on Doppler
* Tributary vein depth > 4 mm from the skin surface
* Pregnancy or breastfeeding
* Known allergy or hypersensitivity to polidocanol
* History of deep vein thrombosis or pulmonary embolism in the last 6 months
* Use of anticoagulant therapy that cannot be safely interrupted
* Active skin infection or ulcer at the treatment site
* Autoimmune or connective tissue disease with active vasculitis
* BMI ≥ 35 kg/m²
* Inability to comply with follow-up visits
* Previous treatment of the target vein in the past 6 months (laser, foam, surgery, or microphlebectomy).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Venous occlusion rate at 30 days | 30 days after the first session
  Ultrasound assessment of the treated vein segment 30 days after the first session, defined as complete absence of detectable flow in the treated vein or partial occlusion with significant reduction in reflux and/or venous diameter, and performed by an independent physician who is blinded to group assignment and not involved in the treatment procedures.

SECONDARY OUTCOMES:
Venous occlusion rate at 90 days | 90 days after the first session
  Ultrasound assessment of the treated vein segment 90 days after the first session, defined as complete occlusion or partial occlusion with improvement inreflux and/or reduction in venous diameter, and performed by an independent physician who is blinded to group assignment and not involved in the treatment procedures.
Final venous occlusion rate at 180 days | 180 days after the first session
  Ultrasound assessment of the treated vein segment 180 days after the first session, defined as complete absence of detectable flow in the treated vein or partial occlusion with significant reduction in reflux and/or venous diameter, and performed by an independent physician who is blinded to group assignment and not involved in the treatment procedures.
Pain intensity immediately after the procedura | Immediately after the procedure (within 30 minutes)
  Participant-reported pain intensity in the treated limb, measured immediately after the session, using a 10-cm Visual Analog Scale (VAS). Higher scores indicate greater pain.
Hyperpigmentation at the treated site | 30, 90, and 180 days after the first session.
  Skin hyperpigmentation will be assessed by an independent physician blinded to the treatment allocation, using standardizes comparative photographs obtained at baseline, 30 days, 90 days, and 180 days.
Number of treatment sessions required | Up to 90 days after the first session.
  Total number of sessions needed to achieve venous occlusion according to the study protocol (maximum of two sessions).
Patient-reported aesthetic satisfaction | Assessed at 90 days after the first session.
  Patient global assessment of cosmetic improvement using a 5-point Likert scale (from "no improvement" to "complete improvement").

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Vieira, PhD, Principal Investigator — Hospital Universitário Pedro Ernesto - UERJ
Locations (1):
- Hospital Universitário Pedro Ernesto - UERJ, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
The study will not share individual particiapnt data (IPD). Aggregate results will be published in scientific journals.